CLINICAL TRIAL: NCT01693523
Title: A Randomized, Placebo Controlled-Double Blind Study of Minocycline for Reducing the Symptom Burden for Pancreatic Cancer Patients
Brief Title: Minocycline Study in Pancreatic Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0587; 1R21CA158902-01A1 (NIH); NCI-2012-02063 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Pancreatic adenocarcinoma; Locally advanced; Metastatic disease; Symptom reduction; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn; Placebo; Sugar Pill; Questionnaires; Surveys
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; cyclopia sequence | interventions — Minocycline; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): Minocycline 100 mg by mouth two times a day (200 mg/day). Initial Dose (starts on first day of run-in phase or chemotherapy). Questionnaires completed at baseline, 1 time each week during drug/placebo administration, and at end of study visit.
  Interventions: Drug: Minocycline; Behavioral: Questionnaires
- Placebo (Placebo Comparator): Matching placebo capsules by mouth twice a day. Initial Dose (starts on first day of run-in phase or chemotherapy). Questionnaires completed at baseline, 1 time each week during drug/placebo administration, and at end of study visit.
  Interventions: Other: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Minocycline — 100 mg by mouth two times a day (200 mg/day).
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Minocycline
Other: Placebo — Matching placebo capsules by mouth twice a day.
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Questionnaires — Questionnaires completed at baseline, 1 time each week during drug/placebo administration, and at end of study visit.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if minocycline can reduce the side effects of chemotherapy in patients with pancreatic cancer. In this study, minocycline will be compared to a placebo.

Minocycline is an antibiotic that may help to reduce side effects of chemotherapy.

A placebo is not a drug. It looks like the study drug, but it is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being in either group:

* If you are in Group 1, you will take minocycline.
* If you are in Group 2, you will take a placebo.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

Each study cycle is about 2 weeks.

You will begin taking the study drug/placebo on, or within 2 days of, Day 1 of the first chemotherapy cycle after you are enrolled on the study. You will take the study drug/placebo capsule by mouth, every day for up to 4 cycles (up to 8 weeks, if there are no treatment delays).

It is possible that your chemotherapy start may be delayed if it takes additional time for your central venous catheter (CVC) to be placed. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. If this happens, you may choose to start taking the study drug/placebo up to 2 weeks before you start chemotherapy, instead of waiting to start taking it on the same day your chemotherapy begins. You can discuss these options with the study doctor.

You should take the study drug/placebo dissolved in a full glass (8 ounces) of water. You may take it with or without food, but if it causes an upset stomach, you should take it with food.

If you have trouble swallowing the dose of study drug/placebo, you can open the capsule right before you take it. You should not lie down for at least 30 minutes after taking the study drug/placebo to reduce the risk of side effects.

You must bring the study drug/placebo container (along with any remaining drug/placebo) to every study visit.

Study Visits:

Before you start your treatment with the study drug/placebo:

* If you can become pregnant, blood (about 2 teaspoons) will be drawn for a pregnancy test. If the pregnancy test is positive, it will be repeated after 48 hours to make sure you are pregnant. Sometimes, cancer can cause a "false positive" on a pregnancy test.
* You will complete 2 questionnaires about pain and other symptoms, and your quality of life. It should take about 5-8 minutes to complete all of the questionnaires.
* If possible, blood (about 2 tablespoons) will be drawn to test for markers of inflammation. Markers of inflammation are found in the blood and may be related to your symptom development.
* Your demographic information, such as your marital status, job status, education, and race will be recorded.

Before you start your chemotherapy treatment:

°If possible, blood (about 2 teaspoons) may be drawn to test for markers of inflammation, only if you started treatment with the study drug/placebo while you waited for your CVC to be placed for chemotherapy. If you choose to wait to start the study drug/placebo until chemotherapy begins, this blood sample will not be drawn.

During treatment with the study drug/placebo:

* You will complete the symptom questionnaire 2 times each week during the first cycle and 1 time each week during any remaining cycles. The symptom questionnaire asks about any symptoms you may be having and how they may be affecting your daily activities. You will also complete the quality of life questionnaire. The questionnaires should take about 3-5 minutes to complete each time.
* You will complete the questionnaires in paper-and-pencil format or on an electronic tablet PC if you are in the clinic. When you are away from the clinic you will complete the questionnaires on the telephone or on your computer.
* If possible, during your clinic visits at the start of cycle 2, 3, and 4 (if applicable), blood (about 2 tablespoons) may be drawn to test for markers of inflammation.

At the end of study drug/placebo treatment:

When you have finished taking the study drug/placebo, the study staff will contact you to complete a questionnaire asking you about your opinions of the study drug/placebo. This questionnaire will take about 3-5 minutes to complete.

Length of Study Participation:

You will be on study for up to 8 weeks, if there is no delay in starting your chemotherapy cycles. You will take the study drug/placebo for up to 8 weeks. You will be taken off study early if the disease gets worse, you have intolerable side effects, if you are unable to follow study directions, or the study doctor thinks it is in your best interest.

End-of-Study Visit:

At the end of the last study cycle after you complete the symptom treatment, you will complete questionnaires about pain and other symptoms and your quality of life. It should take about 3-5 minutes to complete the questionnaires. If possible, blood (about 2 tablespoons) may be drawn to test for markers of inflammation.

Follow-Up:

The study staff will call you 30 days after you finish taking the study drug/placebo to ask about any side effects you may be having. This call should last about 5 minutes.

This is an investigational study. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. Using minocycline to try to reduce the side effects of chemotherapy in patients with pancreatic cancer is investigational.

Up to 76 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Minocycline Trial only: Patients with a pathological or clinical diagnosis of pancreatic cancer and beginning or continuing FOLFIRINOX or gemcitabine-based chemotherapy.
2. Observational Arm only: Patients with a pathological or clinical diagnosis of pancreatic cancer and beginning or continuing FOLFIRINOX chemotherapy.
3. Patients > 18 years old.
4. Minocycline Trial only: Patients with ECOG PS = 0-2.
5. Patients who speak English or Spanish (due to MDASI language options, we are only accruing English-speaking or Spanish-speaking patients to the protocol).
6. Patients willing and able to review, understand, and provide written consent before starting therapy.
7. Minocycline Trial only: Patients with adequate renal function according to MD Anderson testing standards (screening cut off for serum creatinine < 2 times the upper limit of normal).
8. Minocycline Trial only: Patients with adequate hepatic function according to MD Anderson testing standards (screening results for total bilirubin must be < 2 times the upper limit of normal; screening results for alanine aminotransferase (ALT) must be < 3 times the upper limit of normal; screening results for aspartate aminotransferase (AST), if available, must be < 3 times the upper limit of normal).

Exclusion Criteria:

1. Minocycline Trial only: Patients who are taking medication or have conditions that potentially preclude use of minocycline, as determined by the treating physician.
2. Patients who are enrolled in other symptom management clinical trials.
3. Minocycline Trial only: Patients who currently have bile duct obstruction or cholelithiasis.
4. Minocycline Trial only: Patients with hypersensitivity to any tetracyclines.
5. Minocycline Trial only: Patients who are pregnant. Pregnancy will be confirmed by negative urine test; patients with a positive urine test will be retested for doubling of HCG 48 hours after the first test, because of beta-HCG's role as a tumor marker. Patients without such a rise will be eligible for the study and will be enrolled at the investigator's discretion.
6. Minocycline Trial only: Patients who are under treatment of warfarin with INR > 1.5.
7. Patients who, in the judgment of the investigator, may be unable to participate in the required study procedures.
8. Minocycline Trial only: Patients who have had prior treatment for pancreatic cancer within the past six months may be excluded at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Fogelman, MD, Principal Investigator — M.D. Anderson Cancer Center; Shelley Wang, MD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: February 20, 2013 to October, 20 2015. All recruitment done at the University of Texas MD Anderson Cancer
Pre-assignment Details: Of the 80 participants enrolled 1 participant were excluded from the study before assignment to groups.
Groups:
- Observational: No Intervention
Period: Overall Study
Arm/Group | Minocycline | Placebo | Observational
Started | 23 | 21 | 35
Completed | 18 | 13 | 27
Not Completed | 5 | 8 | 8
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Death | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Lack of compliance study medication | 1 | 2 | 0
Not completed — Chemotherapy was held | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Observational: Non Intervention
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Observational | Total
Number analyzed (Participants) | 23 | 21 | 35 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 21 | 49
  >=65 years | 10 | 6 | 14 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 15 | 35
  Male | 12 | 12 | 20 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 1 | 8
  Not Hispanic or Latino | 19 | 18 | 33 | 70
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 6 | 11
  White | 20 | 17 | 28 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 35 | 79

OUTCOME MEASURES:

1. Primary Outcome: Average Area Under the Curve (AUC) of Apriori Selected MDASI Symptoms
Description: Each item is rated on a 0 to 10 scale with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imagine or complete interference using the MD Anderson Symptom Inventory (MDASI). It is a measure of symptom burden, which includes symptom severity and how they interfere with daily functioning. For this study, the sub scale is the average of the 5 pre-selected items namely fatigue, pain, disturbed sleep, lack of appetite and drowsiness. This subscale ranges from 0 to 10. The primary outcome is the average of the 70-day area (10 week study) under the curve for the sub scale. AUC ranges from 0 (0*70) to 700 (10*70). To put this into perspective, the average AUC for the placebo group of 200.8 can also be thought of as 2.87 (200.8/70) on a 0 to 10 scale over the 70 day study period. Lower values represent better outcome. Higher values represent worse outcome.
Time Frame: AUC from baseline to 2 weeks
Population: Of the 44 randomized patients, 30 (68% were evaluable for the primary efficacy analysis).
Measure: Mean (Standard Deviation); unit: Units on a scale *days
Arm/Group | Minocycline | Placebo | Observational
Number analyzed (Participants) | 23 | 21 | 35
Units on a scale *days | 51.5 (31.4) | 30.6 (19.9) | 36.2 (18.8)

2. Secondary Outcome: Relationship Between Dynamic Changes in Inflammation Biomarkers and Symptom Outcomes, Controlling for the Grouping Variables (Tumor Markers, Weight Loss), Evidence of Infection, ECOG PS, Age and Gender Examined
Time Frame: 3 weeks
Population: The blood sample collection was an optional procedure for the participants data were not collected.
Arm/Group | Minocycline | Placebo | Observational
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study and the study completion, an average of 2 years,8 months
Description: Adverse Events were not monitored/assessed for participants in the "Observational" Arm/Group.
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/21
Other Adverse Events (participants affected / at risk) | 3/23 | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=23) | Placebo (N=21)
Septic shock (Infections and infestations) | 2 | 0
Sudden cardiopulmonare (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=23) | Placebo (N=21)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weakness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Splenic infiltarion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT01693523/Prot_SAP_000.pdf